CLINICAL TRIAL: NCT05576909
Title: Donafenib Combined With Hepatic Artery Chemoembolization for Perioperative Treatment of Liver Transplantation: a Single-arm Exploratory Study
Brief Title: Donafenib Combined With Hepatic Artery Chemoembolization for Perioperative Treatment of Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPM-HCC-N03
Record Dates: First submitted 2022-08-14; First posted 2022-10-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib (Experimental): Donafenib combine with TACE for downstaging treatment;
  Donafenib for adjuvant therapy.
  Interventions: Drug: Donafenib; Procedure: TACE

INTERVENTIONS:
Drug: Donafenib — 0.2g BID for downstaging treatment;
  0.1g BID for adjuvant therapy
Procedure: TACE — For downstaging treatment

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the combination of donafenib and TACE in the perioperative period of liver transplantation.

DETAILED DESCRIPTION:
This study plans to enroll about 20 patients with hepatocellular carcinoma (HCC) who do not meet the UCSF standard, they will receive donafenib combined with TACE in downstaging period and donafenib only in adjuvant period.

Before the liver transplantation, the safety and efficacy will be evaluated every 3 and 6 weeks, respectively, until liver transplantation or the disease progression that couldn't be treated by TACE.

After transplantation, the safety and efficacy will be evaluated every 6 and 12 weeks, respectively, until intolerable toxicity, recurrence or up to 12 months treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC either by biopsy or according to AASLD criteria;
2. At least one measurable lesion according to mRECIST;
3. The previous palliative TACE treatment did not exceed one time, with an interval of ≥ 6 months; For patients who had received one prior TACE treatment, the treated lession progressed or lipiodol deposition was less than 50%;
4. Child-Pugh class ≤ 7;
5. ECOG Performance Status 0-1;
6. Intrahepatic tumors meet any of the following conditions:

   * Beyond the UCSF standard, no more than 5 intrahepatic tumors with the longest diameters ≤ 10cm, no tumor thrombus in the main portal vein
   * Meet the UCSF standard, but AFP > 1000 ng / ml

Exclusion Criteria:

1. The pathological diagnosis was hepatocellular carcinoma intrahepatic cholangiocarcinoma (HCC-ICC) mixed type or fibrous lamellar hepatocellular carcinoma;
2. There were inferior vena cava cancer thrombus, hepatic vein cancer thrombus, regional lymph node invasion or extrahepatic metastasis;
3. HCC recurred within 2 years after radical resection or ablation;
4. Patients who have received prior liver transplantation, ≥ 2 times of palliative TACE or other palliative local treatment (including HAIC, radiotherapy, etc.), but who have received prior radical hepatectomy, radical ablation and preventive TACE for the purpose of anti-recurrence can be enrolled;
5. Prior or ongoing systemic therapy (including systemic therapeutic drugs under research, excluding antiviral therapy), including but not limited to TKI such as sorafenib, lenvatinib, regofinib, apatinib, and ambrotinib, PD-1 / PD-L1 monoclonal antibody or immunotherapy against PD-1 / PD-L1, etc;
6. There are contraindications to TACE determined by the investigators (e.g., portal vein trunk obstruction without formation of collateral vessels, etc.);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Downstaging success rate | Immediately after downstaging treatment
  Definition of successful downstaging: those who meet the UCSF standard with baseline AFP > 1000 ng/ml need to be reduced to < 500 ng/ml.

SECONDARY OUTCOMES:
Objective response rate before transplantation (ORR) | 1 year
Complete pathological response rate (pCR) | 1 year
Recurrence-free survival (RFS) | 3 years
  Including median RFS, 1, 2, 3-years RFS rate
Overall survival (OS) | 3 years
  Including median OS, 1, 2, 3-years OS rate
Adverse events | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China